CLINICAL TRIAL: NCT02470026
Title: Influences on Noradrenergic Activity for Cognition in Patients With Major Depressive Disorder
Brief Title: Noradrenergic Activity, Cognition and Major Depressive Disorder
Acronym: YohCog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Linn Kuehl, PhD, PhD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KU3106/2-1
Record Dates: First submitted 2015-05-31; First posted 2015-06-12 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder; Early Life Trauma
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Yohimbine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yohimbine-Placebo (Experimental): single low dose treatment with yohimbine on test day 1, placebo on test day 2
  Interventions: Drug: yohimbine; Drug: placebo
- Placebo-Yohimbin (Experimental): placebo on test day 1, single low dose treatment with yohimbine on test day 2
  Interventions: Drug: yohimbine; Drug: placebo

INTERVENTIONS:
Drug: yohimbine — single low dose treatment
Drug: placebo — single control treatment

SUMMARY:
This study investigates influences of nordadrenergic activity on cognition in patients with major depression regarding influences of early life stress.

DETAILED DESCRIPTION:
Stress plays a major role in the development and maintenance of major depression disorder. Indeed, various studies demonstrated maladaptive changes in physiological stress regulation systems of depressive patients, i.e. in the hypothalamus-pituitary-adrenal axis and the locus coeruleus-noradrenergic system. On a central level, changes of the locus coeruleus-noradrenergic system have been demonstrated.This seems to be the case especially in depressive patients with early life traumata. Comparable to the hypothalamus-pituitary-adrenal axis, the locus coeruleus-noradrenergic system influences not only the physiological stress response, but has also central influence with effects on cognitive functions. Indeed, noradrenergic effects on cognitive functions such as attention, learning and memory have been demonstrated in healthy individuals. Even though deficits in cognitive domains are core symptoms of major depression, the relationship of the noradrenergic system and cognitive processes has rarely been investigated so far.

In this project, the investigators will examine noradrenergic influences via administration of the alpha2-receptor blocker yohimbine on cognitive and emotionally relevant processes in depressive patients and controls. Additionally, the investigators will examine the influence of early life traumata on these relationships. Thus, the investigators will examine participants with and without major depression and with and without early life stress.

Results of this study will improve the understanding of cognitive dysfunctions associated with the noradrenergic system in patients with major depression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depression
* experience of early life trauma

Exclusion Criteria:

* severe illness
* Alzheimer´s
* schizophrenia
* bipolar disorder
* control group: - diagnosis of major depression/ experience of early life trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2014-06; Primary Completion 2017-11 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
behavioral responses in two different conditions of noradrenergic stimulation | 2,5 hrs
  reaction times and error scores (computer tasks)
physiological responses in two different conditions of noradrenergic stimulation | 2,5 hrs
  physiological recordings, saliva samples

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany